CLINICAL TRIAL: NCT02914886
Title: Lipoatrophy in Children, Adolescents and Adults With Modern Treatment Modalities: is There a Beneficial Effect of Insulin Glulisine?
Brief Title: Beneficial Effect of Insulin Glulisine by Lipoatrophy and Type 1 Diabetes (LAS)
Acronym: LAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Olga Kordonouri, Prof. Dr. (MD), Kinderkrankenhaus auf der Bult
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-14652
Record Dates: First submitted 2016-07-08; First posted 2016-09-26 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes; Lipoatrophy
Keywords: Diabetes; Lipoatrophy; children; adolescents; adults; insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Lipodystrophy; Diabetes Mellitus | interventions — insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Daily use of insulin Apidra in insulin pump. The dosis will be according to the patient's former dosing scheme.
  Interventions: Drug: Apidra
- Group 2 (Active Comparator): Daily use of current insulin in insulin pump.The dosis will be according to the patient's former dosing scheme.
  Interventions: Drug: current insulin

INTERVENTIONS:
Drug: Apidra — Half of patients with lipoatrophy will be switched randomly to insulin Apidra for 12 months. Any site other than the lipoatrophic site would be used for delivering the insulin for the purpose of this study.
  Other Names: Glulisine
  Arms: Group 1
Drug: current insulin — Half of patients with lipoatrophy will still use their current Insulin for 6 months. After 6 months the current insulin will be switched to insulin Apidra for the next 6 months.
  Other Names: short-acting analog insulin
  Arms: Group 2

SUMMARY:
The purpose of this study is to investigate whether a zinc-free insulin is an effective treatment option for lipoatrophy in patients with type 1 Diabetes (T1D) and insulin pump (CSII, continuous subcutaneous insulin infusion) therapy.

DETAILED DESCRIPTION:
Randomized, controlled, open-label parallel study. Clinical Study Phase IV After being included in the study, subjects are getting an extensive dermatological examination by a pediatric dermatologist familiar with cutaneous complications of T1D, additionally pathological results will be documented by photography and, if necessary, videodermoscopy. Additionally, an evaluation of their lipoatrophic areas using imaging methods like ultrasound (USG) and MRI will be performed. After randomization, half of the included children switch their pump insulin into insulin glulisine (intervention group) for 6 months. The others continue their current treatment (control group) and switch to insulin glulisine 6 months later. Both groups are followed-up until month 12. Hence, after the 4th visit at 6 months, all enrolled patients are on insulin glulisine pumps for a further period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes and documented lipoatrophy at injection sites on CSII treatment
* Age between 6 and 40 years (both inclusive, see rationale for the inclusion of minors above)
* Signed informed consent form from patients or from parents/their guardians if children/youths <18 years
* Patients must be willing to undergo all study procedures

Exclusion Criteria:

* Patients with previous use of insulin glulisine
* Patients requiring corticosteroids as treatment medication. NOTE inhaled corticosteroids are allowed.
* Patients suffering from severe chronic disease other than T1D or genetic disorder (i.e. Down syndrome etc.)
* Pregnant or lactating women
* Patients participating in other device or drug studies
* History of drug or alcohol abuse within the last five years prior to screening
* Anamnestic history of hypersensitivity to the study drugs (or any component of the study drug) or to drugs with similar chemical structures
* History of severe or multiple allergies
* Treatment with any other investigational drug within 3 months prior to screening
* Progressive fatal disease
* History of significant cardiovascular (such as myocardial infarction, stroke, TIA), respiratory, gastrointestinal, hepatic (ALT and/or AST > 3 times the normal reference range), renal (creatinine > 1.1 mg/dl in women and > 1.5 mg/dl in men), neurological, psychiatric and/or hematological disease as judged by the investigator
* Sexually active women of childbearing potential not consistently and correctly practicing birth control by implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomized partner
* Lack of compliance or other similar reason that, according to investigator, precludes satisfactory participation in the study
* Prisoners or subjects who are involuntarily incarcerated

Target Disease Exclusions

* History of T2DM, maturity onset diabetes of young (MODY), pancreatic surgery or chronic pancreatitis
* Any use of oral hypoglycemic agents within 12 months prior to the screening visit
* History of diabetes ketoacidosis (DKA) within 12 weeks prior to the screening visit
* History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 3 months prior to the screening visit
* Frequent episodes of hypoglycemia as defined by more than one episode requiring assistance, emergency care (paramedics or emergency room care) or glucagon therapy, or more than 2 unexplained episodes of symptomatic hypoglycemia within 3 months prior to the screening visit. An unexplained event is defined as an event that cannot be explained by circumstances such as dietary (e.g. missed meal), strenuous exercise, error in insulin dosing, etc.
* Hypoglycemic unawareness
* History of diabetes insipidus
* History of Addison's disease or chronic adrenal insufficiency

Physical and Laboratory Test Findings

* BMI above 35 kg/m2
* RR > 180/110 mm Hg
* Aspartate aminotransferase (AST) > 3X Upper limit of normal (ULN)
* Alanine aminotransferase (ALT) > 3X ULN
* Serum total bilirubin > 3X ULN
* Estimated GFR (eGFR) < 60 ml/min/1.73 m2
* Hemoglobin ≤ 11.0 g/dl (110 g/l) for boys / men; hemoglobin ≤10.0 g/dl (100 g/L) for girls / women.
* Creatine kinase (CK) > 3X ULN
* Positive for hepatitis B surface antigen or anti-hepatitis C virus antibody.
* Abnormal Free T4 Note: abnormal TSH value at screening will be further evaluated for free T4. Subjects with abnormal free T4 values will be excluded. A one-time retest may be allowed, as determined by the Investigator, after a minimum of 6 weeks following the adjustment of thyroid hormone replacement therapy in subject who have had a prior diagnosis of a thyroid disorder and who are currently receiving thyroid replacement therapy. Such cases should be discussed with the Investigator prior to retesting.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Relative thickness as assessed by MRI | at 6 months
  The relative thickness will be used instead of raw data of the MRI measurements as given by the thickness of the most atrophic region related to the thickness of the reference region of the same patient (normal tissue). The change (increase) of the thickness is defined as difference between the relative thicknesses of the same atrophic region (given as percentage of the same reference region) at 6 months and study begin.

SECONDARY OUTCOMES:
Relative thickness as assessed by MRI | at 6 and 12 months
  Change of relative thickness (as defined above) at 6 and 12 months in the control group
Relative thickness as assessed by MRI | at baseline and 12 months
  Change of relative thickness (as defined above) between baseline and 12 months in both arms
Relative thickness as assessed by USG | at 6 months
  The relative thickness will be used as given by the thickness of the most atrophic region related to the thickness of the reference region of the same patient (normal tissue). The change (increase) of the thickness is defined as difference between the relative thicknesses of the same atrophic region (given as percentage of the same reference region) at 6 months between both groups
Relative thickness as assessed by USG | at 6 and 12 months
  The relative thickness will be used as given by the thickness of the most atrophic region related to the thickness of the reference region of the same patient (normal tissue). The change (increase) of the thickness is defined as difference between the relative thicknesses of the same atrophic region (given as percentage of the same reference region) at 6 months and 12 months in the control group
Relative thickness as assessed by USG | at baseline and 12 months
  The relative thickness will be used as given by the thickness of the most atrophic region related to the thickness of the reference region of the same patient (normal tissue). The change (increase) of the thickness is defined as difference between the relative thicknesses of the same atrophic region (given as percentage of the same reference region) between baseline and 12 months in both groups
indicator dermatoses of Diabetes mellitus and associated autoimmune disorders of the skin | at 6 and 12 months
  Comparison of dermatological findings between 6 and 12 months in the control Group. Dermatological outcome measures will consist in the detection and documentation of a) indicator dermatoses of diabetes mellitus (e. g. lipoatrophy, necrobiosis lipoidica, granuloma anulare), b) associated autoimmune disorders of the skin (e. g. vitiligo, lichen sclerosus, lichen ruber) and c) other, concurrent skin disorders such as atopic dermatitis, acne or psoriasis, for example. If available, disease scores such as the SCORAD score for atopic dermatitis or the PASI score for psoriasis vulgaris will be used to document disease activity.
Number of new lipoatrophic areas | at 6 and 12 months
  Occurrence of new lipoatrophic areas in both arms at 6 and 12 months
Glycemic control | at 6 and 12 months
  Change of HbA1c at 6 and 12 months compared to baseline in both groups
Insulin requirements | at 6 and 12 months
  Change of total daily insulin units per kg body weight at 6 and 12 months compared to baseline in both groups
Laboratory findings | at baseline, 6 months and 12 months
  Comparison of laboratory parameters (insulin antibodies, total IgE, specific insulin-IgE) between baseline, 6 months and 12 months
Side effects | within 12 months
  Side-effects of treatment with other insulins and insulin glulisine such as
  * severe hypoglycemia
  * DKA
  * Catheter occlusion
  * SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Olga Kordonouri, MD, Principal Investigator — Kinder- und Jugendkrankenhaus AUF DER BULT

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kordonouri O, Biester T, Weidemann J, Ott H, Remus K, Grothaus J, Pisarek N, Hartmann R, Adolph K, Lange K, Danne T. Lipoatrophy in children, adolescents and adults with insulin pump treatment: Is there a beneficial effect of insulin glulisine? Pediatr Diabetes. 2020 Nov;21(7):1285-1291. doi: 10.1111/pedi.13094. Epub 2020 Aug 19. PMID 32738019